CLINICAL TRIAL: NCT03608969
Title: Prevalence of Orofacial Dysfunction in Cerebral Palsy Patients by Using Nordic Orofacial Test Screening (NOT-S) and Its Association With Oral Health Status and Quality of Life
Brief Title: Orofacial Dysfunction in Cerebral Palsy Patients and Its Association With Oral Health Status and Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-112
Record Dates: First submitted 2018-06-05; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Orofacial dysfunction; Oral Health; Quality of Life
MeSH Terms: conditions — Cerebral Palsy | interventions — Periodontal Index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Study Group: Children with cerebral palsy aged 3-16 years will be evaluated in terms of the orofacial function using the Nordic Orofacial test- screening (NOT-S). Gross Motor Function Classification System (GMFCS), Manual Ability Classification System (MACS) level and Communication Function Scale (CFS) of child will be recorded. Oral health related quality of life will be assessed using the Parental- Caregiver Perceptions Questionnaire. Caries experience will be measured by identifying decayed, missing, and filled teeth for deciduous and permanent teeth (dmft)
  Interventions: Other: NOT-S

INTERVENTIONS:
Other: NOT-S — Participants are assessed for the orofacial function using the Nordic Orofacial test- screening (NOT-S), Gross Motor Function Classification System (GMFCS), Manual Ability Classification System (MACS) and Communication Function Scale (CFS). Oral health related quality of life is assessed using the Parental- Caregiver Perceptions Questionnaire (P-CPQ). Caries experience was measured by identifying decayed, missing, and filled teeth for deciduous and permanent teeth (dmft). Gingival index and type of occlusion will be recorded.
  Other Names: Gross Motor Function Classification System (GMFCS); Manual Ability Classification System (MACS); Communication Function Scale (CFS); The decayed, missing, and filled teeth (DMFT) index; Parental- Caregiver Perceptions Questionnaire (P-CPQ); Simplified Oral Hygiene Index (OHI-S); Gingival index; Type of occlusion

SUMMARY:
The objective of this study is to analyze prevalence of orofacial dysfunction in children with cerebral palsy by using Nordic Orofacial Test screening (NOT-S) and its association with oral health status and quality of life.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of neurodevelopmental conditions characterized by motor disorders, where orofacial functions, such as controlling saliva, talking, and eating are often affected. Impaired eating is associated with poor growth and problems with chewing and swallowing problems may jeopardize respiration. Notably, the most common causes of death in young individuals with CP are secondary respiratory diseases. Hence, dysfunction in the face, tongue, palate and throat, generically termed orofacial dysfunction has a strong impact on health in individuals with CP. From a dental point of view, early examinations for intervention and prevention among children in general (and those with special needs specifically) are strongly recommended by major dental academies. However, because children with CP have multiple medical issues, their dental issues might not receive equal consideration from healthcare providers trying to provide the best comprehensive care. This can create significant morbidity that can further affect the wellbeing of these compromised children and negatively impact their quality of life.

This study will evaluate the relationship among orofacial functions, manual ability, gross motor function and oral health related quality of life (OHRQOL) in parents / caregivers. One hundred child (4-16 years) will be assessed for orofacial function using the Turkish version for the Nordic Orofacial Test-Screening (NOT-S) protocol, which consists of a structured interview and clinical examination. In NOT-S, aspects of orofacial dysfunction are termed domains. Each domain consists of questions or tasks, which are termed items. Each item serves to discriminate between normal function and dysfunction. The domains and items were finally formulated through discussions in the development team. The NOT-S consists of a structured interview, registering everyday orofacial functions, and a basic clinical examination registering intentional sensory-motor control via the cranial nerves. The interview contains six domains: 'Sensory function', 'Breathing', 'Habits', 'Chewing and swallowing', 'Drooling', and 'Dryness of the mouth'. The examination contains six domains: 'Face at rest', 'Nose breathing', 'Facial expression', 'Masticatory muscle and jaw function', 'Oral motor function', and 'Speech'. Each domain comprises one to five items. Each item is rated with 'yes', if the criterion of dysfunction is fulfilled, or 'no', if not fulfilled. If one or more items within a domain are assessed with 'yes', dysfunction is indicated in the domain.

Self-initiated functional ability will be classified according to the expanded and revised version of the Gross Motor Function Classification System (GMFCS) and Manual Ability Classification System (MACS). Both GMFCS and MACS are five-level systems (I-V) in which level I represents minor and level V represents major limitations in function and ability. Caries Status Caries status will be determined by recording the number of decayed (d, D), missing (m,M), and filled (f, F) teeth in the primary and permanent dentition. With the decayed, missing, and filled teeth (DMFT) index for permanent, and DMFT index for primary dentition we will assess the mean dental caries scores for every individual.

Oral hygiene is a basic factor for oral health. Poor oral hygiene leads to dental plaque collections, which with times turns into the calculus as finally can cause gingivitis and periodontal diseases. That is why many studies, also ours, have been carried out focusing on the role of oral hygiene. Some indices have been developed for assessing individual levels of oral health status. In this study, we decided to use Simplified Oral Hygiene Index (OHI-S). The OHI-S differs from the original OHI in the number of the tooth surfaces scored. Instead of 12, there are just six surfaces. The OHI-S has two components, the Debris Index and the Calculus Index. Each of these indexes is based on numerical determinations representing the amount of the debris or calculus found on the tooth surfaces. The six surfaces examined for the OHI-S are selected from four posterior and two anterior teeth.

Oral health related quality of life measures the functional and psychosocial outcomes of oral disorders. It is now generally accepted in the research community that they are essential as clinical indicators when assessing the oral health of individuals and populations, making clinical decisions, and evaluating dental interventions, services, and programs. According to the US Surgeon General, oral disease and conditions can "…undermine self-image and self-esteem, discourage normal social interaction, and cause other health problems and lead to chronic stress and depression as well as incur great financial cost. They may also interfere with vital functions such as breathing, food selection eating, swallowing and speaking, and with activities of daily living such as work, school, and family interactions". People assess their HRQOL by comparing their expectations and experiences. Parental- Caregiver Perceptions Questionnaire (P-CPQ) was developed to measure parental or caregiver perceptions of a child's OHRQOL and the impact of the child's condition on the family.

The objective of this study is to analyze prevalence of orofacial dysfunction in cerebral palsy patients by using NOT-S and its association with OHRQOL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cerebral palsy aged 3-16 who admit Pediatric Rehabilitation outpatient clinics of Department of Physical Therapy and Rehabilitation of Marmara University School of Medicine

Exclusion Criteria:

1. Patients with uncooperative behavior or not able to understand verbal instructions.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with cerebral palsy aged 3-16 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-10 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Nordic Orofacial Test-Screening (NOT-S) | Day 0
  it has 12 domains distributed between two sections. Six domains are based on an interview (sensory function, breathing, habits, chewing and swallowing, drooling and dry mouth) and six based on a clinical evaluation (face at rest, nose breathing, masticatory muscles and jaw function, oral motor function and speech).

SECONDARY OUTCOMES:
Parental- Caregiver Perceptions Questionnaire (P-CPQ) | Day 0
  Assesses oral health related quality of life. There are four domains tested to ascertain oral health quality of life: oral symptoms, functional limitations, emotional well-being and family well-being/parental distress.
Caries Status (the number of decayed (d, D) teeth) in the primary dentition | Day 0
  the number of decayed (d, D) teeth)
Caries Status (the number of decayed (d, D) teeth) in the permanent dentition | Day 0
  the number of decayed (d, D) teeth)
Caries Status (the number of missing (m,M) teeth) in the primary dentition | Day 0
  the number of missing (m,M) teeth
Caries Status (the number of missing (m,M) teeth) in the permanent dentition | Day 0
  the number of missing (m,M) teeth
Caries Status (the number of filled (f, F) teeth) in the primary dentition | Day 0
  the number of filled (f, F) teeth
Caries Status (the number of filled (f, F) teeth) in the permanent dentition | Day 0
  the number of filled (f, F) teeth
Oral Hygiene Debris Index | Day 0
  Oral hygiene Debris Index is based on numerical determinations representing the amount of the debris found on the tooth surfaces.
Oral Hygiene Calculus Index | Day 0
  Oral Hygiene Calculus Index is based on numerical determinations representing the amount of the calculus found on the tooth surfaces.
Gingival status | Day 0
  Gingival status is used for the assessment of the gingival condition and records qualitative changes in the gingiva.
Type of occlusion | Day 0
  it's classified into three categories: Class 1, Class 2 and Class 3. Teeth are aligned in Cusp Fossa relationship with their antagonist teeth. This is noted as "NORMAL" occlusion
Communication Function Classification System (CFCS) | Day 0
  The CFCS is a tool used to classify the everyday communication of an individual with cerebral palsy into one of five levels according to effectiveness of communication
Gross Motor Function Classification System (GMFCS) | Day 0
  a 5-level classification system that describes the gross motor function of children and youth with cerebral palsy on the basis of their self-initiated movement with particular emphasis on sitting, walking, and wheeled mobility
Manual Ability Classification System (MACS) | Day 0
  The ability of children from 4 - 18 years old with cerebral palsy to handle objects in everyday activities can be categorised into 5 levels using MACS.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Tanboğa, Prof.Dr., Study Director — Marmara university Faculty of Dentistry; Evrim Karadağ, prof.Dr., Study Director — Marmara University; lşıl Özgül Kalyoncu, Asst. Prof., Study Director — Marmara University Faculty of Dentistry; Esra Giray, MD, Study Director — Marmara University; Louay Akkash, DDS, Principal Investigator — Marmara university Faculty of Dentistry; MENNATTALLAH ABDELRAHMAN, DDS, Principal Investigator — Marmara university Faculty of Dentistry
Locations (1):
- Marmara University Researcy And Educational Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Cruz M, Jenkins R, Silberberg D. The burden of brain disorders. Science. 2006 Apr 7;312(5770):53. doi: 10.1126/science.312.5770.53b. No abstract available. PMID 16601174
- [Background] Khandaker G, Smithers-Sheedy H, Islam J, Alam M, Jung J, Novak I, Booy R, Jones C, Badawi N, Muhit M. Bangladesh Cerebral Palsy Register (BCPR): a pilot study to develop a national cerebral palsy (CP) register with surveillance of children for CP. BMC Neurol. 2015 Sep 25;15:173. doi: 10.1186/s12883-015-0427-9. PMID 26407723
- [Background] Dougherty NJ. A review of cerebral palsy for the oral health professional. Dent Clin North Am. 2009 Apr;53(2):329-38, x. doi: 10.1016/j.cden.2008.12.001. PMID 19269401
- [Background] El Ashiry EA, Alaki SM, Nouri SM. Oral Health Quality of Life in Children with Cerebral Palsy: Parental Perceptions. J Clin Pediatr Dent. 2016;40(5):375-87. doi: 10.17796/1053-4628-40.5.375. PMID 27617378
- [Background] Briesemeister M, Schmidt KC, Ries LG. Changes in masticatory muscle activity in children with cerebral palsy. J Electromyogr Kinesiol. 2013 Feb;23(1):260-6. doi: 10.1016/j.jelekin.2012.09.002. Epub 2012 Oct 12. PMID 23063911
- [Background] Bakke M, Bergendal B, McAllister A, Sjogreen L, Asten P. Development and evaluation of a comprehensive screening for orofacial dysfunction. Swed Dent J. 2007;31(2):75-84. PMID 17695052
- [Background] Alev ALAÇAM, Arzu Şükran İNCİOĞLU. Turkish version of The Nordic Orofacial Test - Screening (NOT-S)
- [Background] Lundeborg I, McAllister A, Graf J, Ericsson E, Hultcrantz E. Oral motor dysfunction in children with adenotonsillar hypertrophy--effects of surgery. Logoped Phoniatr Vocol. 2009;34(3):111-6. doi: 10.1080/14015430903066937. PMID 19565403
- [Background] Jokovic A, Locker D, Tompson B, Guyatt G. Questionnaire for measuring oral health-related quality of life in eight- to ten-year-old children. Pediatr Dent. 2004 Nov-Dec;26(6):512-8. PMID 15646914
- [Background] Rozier RG, Pahel BT. Patient- and population-reported outcomes in public health dentistry: oral health-related quality of life. Dent Clin North Am. 2008 Apr;52(2):345-65, vi-vii. doi: 10.1016/j.cden.2007.12.002. PMID 18329448
- [Background] Carr AJ, Gibson B, Robinson PG. Measuring quality of life: Is quality of life determined by expectations or experience? BMJ. 2001 May 19;322(7296):1240-3. doi: 10.1136/bmj.322.7296.1240. No abstract available. PMID 11358783
- [Background] Jokovic A, Locker D, Stephens M, Kenny D, Tompson B, Guyatt G. Measuring parental perceptions of child oral health-related quality of life. J Public Health Dent. 2003 Spring;63(2):67-72. doi: 10.1111/j.1752-7325.2003.tb03477.x. PMID 12816135